CLINICAL TRIAL: NCT03515239
Title: Comparative Study Between Unillateral and Bilateral Lumbopelvic Fixation for Spinopelvic Dissociation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Essam Kamal Rashid, Principal Investigator, Assiut University
Other Study IDs: spinopelvic dissociation
Record Dates: First submitted 2018-04-16; First posted 2018-05-03 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Lumbosacral Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: lumbopelvic fixation for spinopelvic dissociation — unilateral and bilateral lumbopelvic fixation for spinopelvic dissociation

SUMMARY:
Lumbopelvic fixation is the treatment opation for spinopelvic dissociation. In our study we will compare unilateral versus bilateral lumbopelvic fixation as regarding functional outcomes by Majeed score along a period of 12vmonths as a primary measure and metal failure,skin condition and nonunion as secondaries.

DETAILED DESCRIPTION:
Traumatic loss of connection between the spine and pelvis can adopt many forms including lumbosacral fracture dislocation and bilateral sacroiliac dislocation. However, the term spinopelvic dissociation refers to a pathological condition in which this dissociation occurs due to the association of a transverse fracture with sagittal fractures in both sacral wings, result-ing in a proximal segment with the vertebral spine and the proximal sacral fragment, which is mechanically separated from a distal segment formed by the pelvic girdle and the rest of the sacrum.

Spinopelvic dissociation is an important entity to recognize because these fractures are almost uniformly unstable with a very narrow set of criteria for conservative management .

The mechanism of injury includes a very high energy trauma with axial compression on the sacrum.

Various options for internal fixation have been proposed, including percutaneous iliosacral screws, transiliac bars, sacral rods, posterior small plates, or vertical stabilization alone .

Some authors have introduced the technique of triangular posterior osteosynthesis (TPO) in the treatment of vertically unstable pelvic fracture..This is a biplanar fixation able to counterbalance the forces on the posterior pelvic ring during unipodal stance, so as to allow early weight-bearing. The stability of fixation could be confirmed by biomechanical testing of human specimens with transforaminal sacral fractures submitted to cyclic loading. The load to failure of the commonly used internal fixation techniques (sacroiliac screw fixation, plating limited to the sacrum) amounted to 60% of the load to failure of triangular stabilizations. In order to perform the triangular osteosynthesis, we used the Click'X system (Synthes, Oberdorf, Switzerland). Pedicle screws were first inserted in the pedicle of L4. Subsequently caudal screws were implanted into the iliac bone, through the posterior-superior-iliac-spine and parallel to the sacroiliac joint. Once the four screws were inserted, reduction was carried out. Connecting rods were inserted and tightened initially only over the proximal pedicle screws of L4.

The pedicle screws were used as ''joysticks'' in order to achieve reduction in the vertical and horizontal direction at this point, the connecting rod was tightened over the distal screws, therefore stabilizing the fracture. In order to obtain stabilization in the horizontal plane a 6-mm rod was inserted as atransversal cross-link between the two longitudinal connecting rods.e used the Click'X system (Synthes, Oberdorf, Switzerland). Pedicle screws were first inserted in the pedicle of L4. Subsequently caudal screws were implanted into the iliac bone, through the posterior-superior-iliac-spine and parallel to the sacroiliac joint. Once the four screws were inserted, reduction was carried out. Connecting rods were inserted and tightened initially only over the proximal pedicle screws of L4.

The pedicle screws were used as ''joysticks'' in order to achieve reduction in the vertical and horizontal direction at this point, the connecting rod was tightened over the distal screws, therefore stabilizing the fracture. In order to obtain stabilization in the horizontal plane a 6-mm rod was inserted as a transversal cross-link between the two longitudinal connecting rods.

ELIGIBILITY:
Inclusion Criteria:

* injury severity score <22
* neurologically free patient

Exclusion Criteria:

* injury severity score >22
* patient with neurological injury

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Skeletally mature and neurologically free patient
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Functional outcomes by Majeed score | Along a period of 12 monthes.
  Functional outcomes by Majeed score in group of patient with spinopelvic dissociation fixed by unilateral triangular osteosynthesis and comparing them with group of patient fixed by bilateral triangular osteosynthesis.

REFERENCES:
- [Background] Denis F, Davis S, Comfort T. Sacral fractures: an important problem. Retrospective analysis of 236 cases. Clin Orthop Relat Res. 1988 Feb;227:67-81. PMID 3338224
- [Background] Roy-Camille R, Saillant G, Gagna G, Mazel C. Transverse fracture of the upper sacrum. Suicidal jumper's fracture. Spine (Phila Pa 1976). 1985 Nov;10(9):838-45. doi: 10.1097/00007632-198511000-00011. PMID 4089659
- [Background] Gibbons KJ, Soloniuk DS, Razack N. Neurological injury and patterns of sacral fractures. J Neurosurg. 1990 Jun;72(6):889-93. doi: 10.3171/jns.1990.72.6.0889. PMID 2338573